CLINICAL TRIAL: NCT02444013
Title: Periprocedural Administration of Folic Acid for Prevention of Contrast Induced Nephropathy in Patients Undergoing Coronary CTA/Angiography/Angioplasty
Brief Title: Folic Acid for Prevention of Contrast Induced Nephropathy
Acronym: FAPCIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinlai Liu, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SYSU-2015
Record Dates: First submitted 2015-04-07; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Diseases; Urologic Diseases
Keywords: Contrast induced nephropathy
MeSH Terms: conditions — Kidney Diseases; Urologic Diseases | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folic acid (Active Comparator): Oral folic acid (5 mg, tid) were given at least two days before CTA/angiography/angioplasty and continued for two days after.
  Interventions: Drug: Folic acid
- Placebo (Placebo Comparator): Oral placebo (1 tablet, tid) were given at least two days before CTA/angiography/angioplasty and continued for two days after.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folic acid
  Other Names: Folic uric acid
  Arms: Folic acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether periprocedural administration of folic acid is effective in the prevention of contrast induced nephropathy in patients undergoing coronary CTA/angiography/angioplasty.

DETAILED DESCRIPTION:
Hyperhomocysteinemia is considered to be independently associated with a greater risk of contrast induced nephropathy (CIN) in previous studies. However, the relationship between homocysteine-lowering therapy and CIN remains uncertain. Folic acid is considered to be the most common agent for homocysteine-lowering therapy. Therefore, this study aims to determine whether periprocedural administration of folic acid is effective in the prevention of CIN. 400 patients undergoing coronary CTA/angiography/angioplasty are going to be initially enrolled. Of these patients,200 were randomly assigned to receive a standard dose of folic acid (5mg tid, given at least two days before the procedural and continued for two days after), 200 to receive placebo. Blood samples for estimations of serum creatinine were collected at 0, 24 and 48h of contrast agent administration. CIN is defined as an elevation of creatinine by ≥ 25% or ≥ 0.5 mg/dl from baseline within 48h. The occurrence of CIN and the major in-hospital clinical events were recorded and compared between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients undergoing coronary CTA/angiography/angioplasty

Exclusion Criteria:

* exposure to nephrotoxic drugs prior to or during the study period
* end-stage renal failure requiring dialysis
* allergy to iodine-containing contrast medium
* pregnancy
* refusal to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of contrast-induced nephropathy | Within 48 hours after contrast exposure
  Contrast-induced nephropathy is defined as an elevation of serum creatinine of more than 25% or ≥0.5 mg/dl (44 μmol/l) from baseline within 48 hours after contrast exposure

SECONDARY OUTCOMES:
Major in-hospital clinical events, including death and need for dialysis or hemofiltration | participants will be followed for the duration of hospital stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jinlai Liu, M.D., Principal Investigator — Organizational Affiliation
Locations (1):
- Department of Cardiology, the Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Kim SJ, Choi D, Ko YG, Kim JS, Han SH, Kim BK, Kang SW, Hong MK, Jang Y, Choi KH, Yoo TH. Relation of homocysteinemia to contrast-induced nephropathy in patients undergoing percutaneous coronary intervention. Am J Cardiol. 2011 Oct 15;108(8):1086-91. doi: 10.1016/j.amjcard.2011.06.010. Epub 2011 Jul 24. PMID 21791335
- [Background] Barbieri L, Verdoia M, Schaffer A, Niccoli G, Perrone-Filardi P, Bellomo G, Marino P, Suryapranata H, Luca GD. Elevated homocysteine and the risk of contrast-induced nephropathy: a cohort study. Angiology. 2015 Apr;66(4):333-8. doi: 10.1177/0003319714533401. Epub 2014 May 15. PMID 24830422
- [Background] Li S, Tang X, Peng L, Luo Y, Zhao Y, Chen L, Dong R, Zhu J, Chen Y, Liu J. A head-to-head comparison of homocysteine and cystatin C as pre-procedure predictors for contrast-induced nephropathy in patients undergoing coronary computed tomography angiography. Clin Chim Acta. 2015 Apr 15;444:86-91. doi: 10.1016/j.cca.2015.02.019. Epub 2015 Feb 14. PMID 25687162
- [Derived] Peng L, Shui X, Tan F, Li Z, Ling Y, Wu B, Chen L, Li S, Peng H. Folic Acid Attenuates Contrast-Induced Nephropathy in Patients With Hyperhomocysteinemia Undergoing Coronary Catheterization: A Randomized Controlled Trial. Front Cardiovasc Med. 2021 Oct 1;8:707328. doi: 10.3389/fcvm.2021.707328. eCollection 2021. PMID 34660712